CLINICAL TRIAL: NCT05196399
Title: A Single-center, Open-label, Randomized, Two-way Crossover Phase 1 Study to Compare the Single-dose Pharmacokinetics of Different Tablet Formulations of Aprocitentan in Healthy Subjects
Brief Title: Bioequivalence Study of Different Aprocitentan Tablet Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ID-080-110; 2021-005090-11 (EudraCT Number)
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — aprocitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aprocitentan (reference product) (Experimental): 25 mg film-coated tablet
  Interventions: Drug: Aprocitentan (Formulation A)
- Aprocitentan (test product) (Experimental): 25 mg film-coated tablet
  Interventions: Drug: Aprocitentan (Formulation B)

INTERVENTIONS:
Drug: Aprocitentan (Formulation A) — A single oral dose of 25 mg.
  Other Names: ACT-132577
  Arms: Aprocitentan (reference product)
Drug: Aprocitentan (Formulation B) — A single oral dose of 25 mg.
  Other Names: ACT-132577
  Arms: Aprocitentan (test product)

SUMMARY:
The main purpose is to study the pharmacokinetics of aprocitentan (ACT-132577) using 2 different tablet formulations. The clinical pharmacology data will be used to determine bioequivalence of 2 different tablet formulations.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Healthy male or female participant aged between 18 and 55 years (inclusive) at Screening.
* Body Mass Index of 18.0 to 30.0 kg/m2 (inclusive) at Screening.
* Systolic blood pressure (SBP) 100-140 mmHg, Diastolic blood pressure (DBP) 60-90 mmHg, and pulse rate 60-100 bpm (inclusive), measured on the dominant arm, after 5 min in the supine position at Screening and on Day 1 pre-dose of the first period.
* Woman of Childbearing Potential who has a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1 of the first period. She must agree to consistently and correctly use (from Screening, during the entire study, and for at least 30 days after the last study treatment administration) a highly effective method of contraception with a failure rate of less than 1% per year.
* Woman of non-childbearing potential, i.e., postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause; in addition, an FSH test must be performed at Screening to further support postmenopausal status), with previous bilateral salpingectomy, bilateral salpingo oophorectomy or hysterectomy, or with premature ovarian failure (confirmed by a specialist), XY genotype, uterine agenesis.

Exclusion Criteria:

* Pregnant or lactating woman.
* Previous administration of aprocitentan.
* Known hypersensitivity to endothelin receptor antagonists or to excipients used in any of the formulations.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatments (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the study results.
* Clinically relevant findings on the physical examination at Screening and on Day -1 of the first period.
* Clinically relevant findings in clinical laboratory tests (hematology and clinical chemistry) at Screening and on Day -1 of the first period.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 3 weeks or 5 terminal elimination half-lives (t½; whichever is longer) prior to first study treatment administration.
* Legal incapacity or limited legal capacity at Screening.
* Positive COVID-19 test, if performed (subject to current epidemiological regulations in the Czech Republic) during the screening period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of aprocitentan | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 10.
The area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification (AUC0-t) of aprocitentan | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 10.
Area under the plasma concentration-time curve from zero to infinity (AUC0-inf) of aprocitentan | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 10.

SECONDARY OUTCOMES:
Treatment-emergent adverse events | From study treatment administration on Day 1 up to last assessment at End of Period (Day 10).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No